CLINICAL TRIAL: NCT07065617
Title: A Phase I, Open-label, Two-part Trial to Investigate the Mass Balance, Metabolism, and Basic Pharmacokinetics of BI 1819479 (C-14) Administered as an Oral Solution (Part A) and to Investigate the Absolute Bioavailability of BI 1819479 Administered as a Film-coated Tablet Together With an Intravenous Microtracer Dose of [14 C]BI 1819479 (Part B) in Healthy Male Volunteers
Brief Title: A Study to Test How BI 1819479 is Taken up and Processed by the Body
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1462-0007
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Healthy
MeSH Terms: interventions — Carbon-14

STUDY DESIGN:
Intervention Model Description: Part A is a single arm trial whereas Part B is conducted in a fixed-sequence.
Masking Description: Both parts are conducted open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: BI 1819479 (C-14) (Experimental)
  Interventions: Drug: BI 1819479 (C-14)
- Part B: BI 1819479, then [14C]BI 1819479 (Experimental)
  Interventions: Drug: [14C]BI 1819479; Drug: BI 1819479

INTERVENTIONS:
Drug: [14C]BI 1819479 — [14C]BI 1819479
  Arms: Part B: BI 1819479, then [14C]BI 1819479
Drug: BI 1819479 — BI 1819479
  Arms: Part B: BI 1819479, then [14C]BI 1819479
Drug: BI 1819479 (C-14) — BI 1819479 mixed with [14C]BI 1819479
  Arms: Part A: BI 1819479 (C-14)

SUMMARY:
This trial is intended to investigate the mass balance, metabolism, and basic pharmacokinetics of BI 1819479 (C-14) (Part A) and to investigate the absolute bioavailability of BI 1819479 (Part B) in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male participants according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests without any clinically significant abnormalities
2. Age of 18 to 55 years (inclusive)
3. Body Mass Index (BMI) of 18.5 to 32.0 kg/m^2 (inclusive)
4. Signed and dated written informed consent in accordance with International Conference of Harmonization-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
5. Must have regular bowel movements (i.e. average stool production of ≥1 and ≤3 stools per day), applicable to Part A only

Exclusion Criteria:

1. Any finding in the medical examination (including vital signs or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 40 to 90 mm Hg, or heart rate outside the range of 45 to 90 bpm (beats per minute)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders, assessed as clinically relevant by the investigator
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2025-08-04 (Actual); Primary Completion 2025-10-04 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Part A: fraction of [14C]-radioactivity excreted in urine as percentage of the administered dose over the time interval from 0 to the last quantifiable time point (fe urine, 0-tz) | Up to 37 days.
Part A: fraction of [14C]-radioactivity excreted in urine as percentage of the administered dose over the time interval from 0 to the last quantifiable time point (fe faeces, 0-tz) | Up to 37 days.
Part B: area under the concentration-time curve of [14C]BI 1819479 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 31 days.

SECONDARY OUTCOMES:
Part A: Maximum measured concentration of [14C]BI 1819479-EQ in plasma (Cmax) | Up to 36 days.
Part A: Area under the concentration-time curve of [14C]BI 1819479-EQ in plasma over the time interval from 0 to the last quantifiable data point (AUC 0-tz) | Up to 36 days.
Part B: Maximum measured concentration of [14C]BI 1819479 in plasma (Cmax) | Up to 31 days.
Part B: Maximum measured concentration of BI 1819479 in plasma (Cmax) | Up to 31 days.
Part B: Area under the concentration-time curve of [14C]BI 1819479 in plasma over the time interval from 0 to the last quantifiable data point (AUC 0-tz) | Up to 31 days.
Part B: Area under the concentration-time curve of BI 1819479 in plasma over the time interval from 0 to the last quantifiable data point (AUC 0-tz) | Up to 31 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com